CLINICAL TRIAL: NCT02127866
Title: A MULTICENTRE, RANDOMISED, DOUBLE-BLIND, ACTIVE-CONTROLLED, 3-WAY CROSS-OVER STUDY TO EVALUATE THE EFFICACY AND SAFETY OF A FREE COMBINATION OF 3 DOSES OF CHF 5259 (GLYCOPYRROLATE) PLUS FOSTER® 100/6 µg (FIXED COMBINATION OF BECLOMETHASONE DIPROPIONATE PLUS FORMOTEROL) IN A METERED DOSE INHALER FOR THE TREATMENT OF PATIENTS WITH UNCONTROLLED ASTHMA UNDER MEDIUM DOSES OF INHALED CORTICOSTEROIDS PLUS LONG-ACTING β2-AGONISTS
Brief Title: Triple in Asthma Dose Finding
Acronym: Triskel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-1206-PR-0088; 2013-003043-36 (EudraCT Number)
Record Dates: First submitted 2014-04-09; First posted 2014-05-01 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Asthma
Keywords: Asthma, anticholinergics
MeSH Terms: conditions — Asthma | interventions — Foster Home Care; Glycopyrrolate; Beclomethasone; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- CHF 5259 25 µg plus Foster 100/6 µg (Experimental)
  Interventions: Drug: CHF 5259 plus Foster 100/6 µg
- CHF 5259 50 µg plus Foster 100/6 µg (Experimental)
  Interventions: Drug: CHF 5259 plus Foster 100/6 µg
- CHF 5259 100 µg plus Foster 100/6 µg (Experimental)
  Interventions: Drug: CHF 5259 plus Foster 100/6 µg
- Foster 100/6 µg (Active Comparator)
  Interventions: Drug: Foster 100/6 µg

INTERVENTIONS:
Drug: CHF 5259 plus Foster 100/6 µg — Comparison of different doses of CHF 5259 (on top of Foster 100 /6 µg) versus Foster 100/6 µg over a treatment period of 6 weeks. Each subject will be allocated to 3 ouf of the 4 possible treatments performed in sequence during a cross over design (incomplete block)
  Other Names: glycopyrrolate + beclometasone/formoterol
  Arms: CHF 5259 100 µg plus Foster 100/6 µg; CHF 5259 25 µg plus Foster 100/6 µg; CHF 5259 50 µg plus Foster 100/6 µg
Drug: Foster 100/6 µg — Active comparator
  Comparison of different doses of CHF 5259 (on top of Foster 100 /6 µg) versus Foster 100/6 µg over a treatment period of 6 weeks. Each subject will be allocated to 3 ouf of the 4 possible treatments performed in sequence during a cross over design (incomplete block)
  Other Names: beclometasone dipropionate/formoterol
  Arms: Foster 100/6 µg

SUMMARY:
The purpose of this study is to determine the optimal dose of CHF 5259 (glycopyrrolate bromide) on top of Foster which provides the optimal additive bronchodilator effect to asthmatic patients whose symptoms are uncontrolled with medium dose of inhaled corticosteroids plus long acting beta2 agonists.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged >=18 years
* Uncontrolled asthma on medium doses of ICS+LABA with ACQ >=1.5
* Pre-bronchodilator FEV1 ≥40% and <80% of their predicted normal value

Exclusion Criteria:

* Pregnant or lactating women
* Diagnosis of COPD
* Patients treated for asthma exacerbations in the 4 weeks prior to study entry
* Patients who are in therapy for gastroesophageal reflux disease
* Patients who have a clinically significant cardiovascular condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
FEV1 AUC0-12h normalised by time on Day 42 | Day 42

SECONDARY OUTCOMES:
Peak FEV1 on Day 42 | Day 42
Adverse Events and Adverse Drug Reactions | Up at Week 24 (study end)

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, MD, Principal Investigator — University Hospital of South Manchester, MANCHESTER M23 9 QZ, UK
Locations (44):
- Bulgaria (10):
  - Chiesi Clinical Trial Site 0105, Dupnitsa
  - Chiesi Clinical Trial Site 0101, Rousse
  - Chiesi Clinical Trial Site 0106, Sevlievo
  - Chiesi Clinical Trial Site 0107, Sofia
  - Chiesi Clinical Trial Site 0108, Sofia
  - Chiesi Clinical Trial Site 0102, Sofia
  - Chiesi Clinical Trial Site 0110, Sofia
  - Chiesi Clinical Trial Site 0109, Sofia
  - Chiesi Clinical Trial Site 0103, Stara Zagora
  - Chiesi Clinical Trial Site 0104, Troyan Municipality
- Germany (8):
  - Chiesi Clinical Trial Site 0208, Berlin
  - Chiesi Clinical Trial Site 0207, Berlin
  - Chiesi Clinical Trial Site 0206, Großhansdorf
  - Chiesi Clinical Trial Site 0201, Leipzig
  - Chiesi Clinical Trial Site 0203, Lübeck
  - Chiesi Clinical Trial Site 0202, Magdeburg
  - Chiesi Clinical Trial Site 0204, Radebeul
  - Chiesi Clinical Trial Site 0210, Witten
- Hungary (7):
  - Chiesi Clinical Trial Site 0307, Balassagyarmat
  - Chiesi Clinical Trial Site 0302, Budapest
  - Chiesi Clinical Trial Site 0304, Deszk
  - Chiesi Clinical Trial Site 0305, Gödöllő
  - Chiesi Clinical Trial Site 0303, Komárom
  - Chiesi Clinical Trial Site 0301, Siófok
  - Chiesi Clinical Trial Site 0306, Szarvas
- Italy (5):
  - Chiesi Clinical Trial Site 0403, Brescia
  - Chiesi Clinical Trial Site 0402, Parma
  - Chiesi Clinical Trial Site 0401, Pisa
  - Chiesi Clinical Trial Site 0408, Trieste
  - Chiesi Clinical Trial Site 0404, Verona
- Poland (12):
  - Chiesi Clinical Trial Site 0510, Bialystok
  - Chiesi Clinical Trial Site 0507, Gdansk
  - Chiesi Clinical Trial Site 0502, Giżycko
  - Chiesi Clinical Trial Site 0511, Krakow
  - Chiesi Clinical Trial Site 0505, Lodz
  - Chiesi Clinical Trial Site 0509, Lodz
  - Chiesi Clinical Trial Site 0512, Lublin
  - Chiesi Clinical Trial Site 0503, Ostróda
  - Chiesi Clinical Trial Site 0501, Oświęcim
  - Chiesi Clinical Trial Site 0506, Proszowice
  - Chiesi Clinical Trial Site 0508, Rzeszów
  - Chiesi Clinical Trial Site 0504, Wroclaw
- United Kingdom (2):
  - Chiesi Clinical Trial Site 0602, London
  - Chiesi Clinical Trial Site 0601, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Chiesi commits to sharing with qualified scientific and medical Researchers, conducting legitimate research, Patient-level Data, Study-level Data, the Clinical Protocol and the full CSR, providing access to clinical trial information consistently with the principle of safeguarding commercially confidential information and patient privacy. Any shared Patient-level Data is anonymized to protect personally identifiable information.
  Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
Access Criteria: Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
URL: https://www.chiesi.com/en/chiesi-clinical-trial-data-request-portal/

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2013-003043-36